CLINICAL TRIAL: NCT05269355
Title: A Phase 2/3 Study to Evaluate the Efficacy and Safety of Unesbulin in Unresectable or Metastatic, Relapsed or Refractory Leiomyosarcoma
Brief Title: A Study of Unesbulin in Participants With Advanced Leiomyosarcoma (LMS)
Acronym: SUNRISELMS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTC596-ONC-008-LMS; 2022-000073-12 (EudraCT Number)
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — PTC596; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Unesbulin and Dacarbazine (Experimental): Participants will receive unesbulin 300 milligrams (mg) tablets administered orally twice weekly in each 3-week treatment cycle in combination with dacarbazine 1000 mg/meter squared (m^2) intravenously (IV) once every 21 days. Treatment will continue for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
  Interventions: Drug: Unesbulin; Drug: Dacarbazine
- Placebo and Dacarbazine (Placebo Comparator): Participants will receive placebo matching to unesbulin tablets administered orally twice weekly in each 3-week treatment cycle in combination with dacarbazine 1000 mg/m^2 IV once every 21 days. Treatment will continue for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
  Interventions: Drug: Dacarbazine; Other: Placebo

INTERVENTIONS:
Drug: Unesbulin — Unesbulin will be administered as per the dose and schedule specified in the arm description.
  Other Names: PTC596
  Arms: Unesbulin and Dacarbazine
Drug: Dacarbazine — Dacarbazine will be administered as per the dose and schedule specified in the arm description.
  Other Names: DTIC
Other: Placebo — Placebo will be administered as per the schedule specified in the arm description.
  Arms: Placebo and Dacarbazine

SUMMARY:
This study will compare the efficacy and safety of unesbulin plus dacarbazine versus placebo plus dacarbazine in participants with unresectable or metastatic, relapsed or refractory LMS who have received at least 1 prior line of systemic therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Histological or cytological confirmation of LMS arising at any anatomic site except bone sarcoma, unresectable or metastatic, relapsed or refractory disease measurable per RECIST 1.1 criteria
* Disease progression on previous treatment before screening or intolerability to other oncology treatments
* Participants with liver metastases may be enrolled
* Participants with well-controlled asthma or chronic obstructive pulmonary disease may be enrolled.
* Toxicity from prior therapies recovered to Grade ≤1 or participant's baseline, except for alopecia. In addition, endocrinopathies associated with prior immunotherapy-based treatments that are well controlled on replacement medication are not exclusionary.
* At least 1 prior systemic cytotoxic or targeted therapy regimen for LMS, which may include but is not limited to single-agent doxorubicin or other anthracycline, doxorubicin plus ifosfamide, trabectedin, pazopanib, or gemcitabine with or without docetaxel.
* At least 4 weeks since prior surgery and recovered in the opinion of investigator

Key Exclusion Criteria:

* Received temozolomide or dacarbazine at any time
* Any other systemic anticancer therapy including investigational agents ≤3 weeks before initiation of study treatment. Additionally, participants may not have received radiation ≤3 weeks before initiation of study treatment.
* Known intolerance to dacarbazine or one or more of the excipients in unesbulin.
* Co-existing active infection or any co-existing medical condition likely to interfere with study procedures
* Gastrointestinal disease or other conditions that could affect absorption. Active peptic ulcer disease, active gastritis, or previous history of gastric perforation within the last 2 years
* Major surgery, open biopsy, or significant traumatic injury that has not recovered, in the opinion of the investigator, within 28 days of baseline
* Immunization with a live vaccine within 30 days before starting study drug due to the risk of serious and life-threatening infections.
* Prior malignancies, other than LMS, that required treatment or have shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ, prostate cancer in situ or any other low risk malignancy that is approved by the medical monitor) during the 5 years before initiation.
* Prior or ongoing clinically significant illness, medical or psychiatric condition, medical history, physical findings, electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant, or alter the absorption, distribution, metabolism, or excretion of the study drugs, or could impair the assessment of study results.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rance, MD, Study Director — PTC Therapeutics
Locations (54):
- United States (23):
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA) - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - University of Florida (UF) Health Cancer Center - Orlando Health, Orlando, Florida
  - Moffitt, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern Medicine - Warrenville Cancer Center, Warrenville, Illinois
  - Johns Hopkins Oncology Group, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - The Trustees of Columbia University, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University (OSU), Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown
  - Peter MacCallum Cancer Institute, East Melbourne
  - Prince of Wales Hospital, Randwick
- Brazil (6):
  - Fundacao PIO XII - Hospital de Amor, Barretos
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - INCA I - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital Sao Rafael - Instituto D'Or da Bahia, Salvador
  - CIP - Centro Integrado de Pesquisas do Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
  - Instituto do Cancer do Estado de São Paulo (ICESP), São Paulo
- Canada (3):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont (HMR), Montreal, Quebec
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsmedizin Mannheim, Mannheim
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
- Eszak-Pesti Centrumkorhaz - Honvedkorhaz, Budapest, Hungary
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - La Fondazione e l'Istituto di Candiolo, Torino
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (2):
  - Niepubliczny Zaklad Opieki Zdrowotnej Zespól Poradni Specjalistycznych "TERMEDICA", Poznan
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- Spain (4):
  - Institut Catala d'Oncologia (Hospital Duran y Reynals), Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - Beatson, West of Scotland Cancer Centre, Glasgow
  - Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 2:1 to 1 of the following treatment groups: 1. Unesbulin and Dacarbazine or 2. Placebo and Dacarbazine.
Groups:
- Unesbulin and Dacarbazine: Participants received unesbulin 300 milligrams (mg) tablets administered orally twice weekly in each 3-week treatment cycle in combination with dacarbazine 1000 mg/square meter (m^2) intravenously (IV) once every 21 days. Treatment was continued for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
- Placebo and Dacarbazine: Participants received placebo matching to unesbulin tablets administered orally twice weekly in each 3-week treatment cycle in combination with dacarbazine 1000 mg/m^2 IV once every 21 days. Treatment was continued for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
Period: Overall Study
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Started | 239 | 120
Received at Least 1 Dose of Study Drug | 238 | 120
Completed | 0 | 0
Not Completed | 239 | 120
Not completed — Progressive Disease | 104 | 68
Not completed — Study Terminated by Sponsor | 87 | 29
Not completed — Adverse Event | 15 | 8
Not completed — Withdrawal by Subject | 18 | 5
Not completed — Physician Decision | 6 | 4
Not completed — Death | 3 | 5
Not completed — Other Than Specified | 5 | 1
Not completed — Randomized But Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug (unesbulin/placebo or dacarbazine).
Groups:
- Unesbulin and Dacarbazine: Participants received unesbulin 300 mg tablets administered orally twice weekly in each 3-week treatment cycle in combination with dacarbazine 1000 mg/m^2 IV once every 21 days. Treatment was continued for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
- Total: Total of all reporting groups
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine | Total
Number analyzed (Participants) | 238 | 120 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.98) | 58.6 (11.04) | 57.8 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 93 | 280
  Male | 51 | 27 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 26 | 62
  Not Hispanic or Latino | 170 | 87 | 257
  Unknown or Not Reported | 32 | 7 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 17 | 8 | 25
  Race: American Indian/Alaska Native | 0 | 1 | 1
  Race: Black/African American | 20 | 6 | 26
  Race: Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
  Race: White/Caucasian | 157 | 92 | 249
  Race: Other | 38 | 12 | 50
  Race: Missing | 2 | 1 | 3
  Race: Multiple | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Independent Central Review Using Response Evaluation Criteria in Solid Tumors (RECIST) V1.1
Description: PFS was defined as the time from randomization to the documented disease progression or death due to any cause, whichever occurred first. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions was also considered progression.
Time Frame: Up to approximately 2 years
Population: The modified intent-to-treat (mITT) set included randomized participants with 1 to 3 prior lines of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 209 | 105
months | 3.6 [2.8 to 5.5] | 2.6 [1.5 to 3.0]
Statistical Analysis 1: Comparison: Unesbulin and Dacarbazine vs Placebo and Dacarbazine; Test type: Other; p = 0.0017, Regression, Cox; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.45 to 0.83]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from the randomization date to the date of death from any cause or date last known alive for those who did not die.
Time Frame: Up to approximately 2 years
Population: The mITT set included randomized participants with 1 to 3 prior lines of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 209 | 105
months | NA [10.4 to NA] — Due to limited number of participants with an event, median and upper limit of 95% confidence interval (CI) could not be calculated. | NA [11.0 to NA] — Due to limited number of participants with an event, median and upper limit of 95% CI could not be calculated.

3. Secondary Outcome: Objective Response Rate (ORR) Per Independent Central Review Using RECIST V1.1
Description: ORR was defined as percentage of participants who achieved a confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 2 years
Population: The mITT set included randomized participants with 1 to 3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 209 | 105
percentage of participants | 8.1 [4.7 to 12.8] | 2.1 [0.3 to 7.3]

4. Secondary Outcome: Disease Control Rate (DCR) Per Independent Central Review Using RECIST V1.1
Description: DCR was defined as percentage of participants who achieved a confirmed BOR of CR, PR, or at least 3 months of stable disease (SD). CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to approximately 2 years
Population: The mITT set included randomized participants with 1 to 3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 209 | 105
percentage of participants | 36.4 [29.7 to 43.5] | 27.1 [18.5 to 37.1]

5. Secondary Outcome: Duration of Response Per Independent Central Review Using RECIST V1.1
Description: Duration of response was defined as the time from the date of first confirmed response of CR or PR to the date of the first documented disease progression or death due to any cause, whichever occurred first. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: Up to approximately 2 years
Population: The mITT set included randomized participants with 1 to 3 prior lines of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 209 | 105
months | 6.87 [NA to NA] — Due to limited number of participants with an event, upper and lower limit of 95% CI could not be calculated. | NA [NA to NA] — Due to limited number of participants with an event, median and upper and lower limit of 95% CI could not be calculated.

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A TEAE was defined as an AE that had an onset date on or after the first dose of study drug until 30 days after last dose or occurred prior to first dose of study drug and worsened in severity after first dose of study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first dose of study drug up to approximately 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 238 | 120
Participants | 236 | 112

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 2 years
Description: The safety analysis set included all participants who received at least 1 dose of study drug (unesbulin/placebo or dacarbazine).
Arm/Group | Unesbulin and Dacarbazine | Placebo and Dacarbazine
All-Cause Mortality (participants affected / at risk) | 49/238 | 27/120
Serious Adverse Events (participants affected / at risk) | 81/238 | 43/120
Other Adverse Events (participants affected / at risk) | 234/238 | 112/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Unesbulin and Dacarbazine (N=238) | Placebo and Dacarbazine (N=120)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 3 | 5
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 5
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 5 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 1
Spinal cord infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 5 | 1
Transaminases increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 1
Device occlusion (Product Issues) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/187 | 0/93 — This is a sex-specific AE. Only female participants were at risk.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Unesbulin and Dacarbazine (N=238) | Placebo and Dacarbazine (N=120)
Anaemia (Blood and lymphatic system disorders) | 103 | 35
Leukopenia (Blood and lymphatic system disorders) | 15 | 7
Neutropenia (Blood and lymphatic system disorders) | 88 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 75 | 27
Abdominal pain (Gastrointestinal disorders) | 42 | 11
Abdominal pain upper (Gastrointestinal disorders) | 13 | 6
Constipation (Gastrointestinal disorders) | 50 | 19
Diarrhoea (Gastrointestinal disorders) | 131 | 27
Nausea (Gastrointestinal disorders) | 115 | 44
Vomiting (Gastrointestinal disorders) | 43 | 17
Asthenia (General disorders) | 27 | 12
Fatigue (General disorders) | 93 | 44
Non-cardiac chest pain (General disorders) | 15 | 5
Oedema peripheral (General disorders) | 20 | 12
Pyrexia (General disorders) | 15 | 9
COVID-19 (Infections and infestations) | 13 | 9
Urinary tract infection (Infections and infestations) | 14 | 8
Alanine aminotransferase increased (Investigations) | 18 | 10
Aspartate aminotransferase increased (Investigations) | 20 | 8
Blood creatinine increased (Investigations) | 13 | 5
Neutrophil count decreased (Investigations) | 60 | 13
Platelet count decreased (Investigations) | 51 | 17
White blood cell count decreased (Investigations) | 36 | 9
Decreased appetite (Metabolism and nutrition disorders) | 37 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 5
Dizziness (Nervous system disorders) | 32 | 10
Dysgeusia (Nervous system disorders) | 17 | 2
Headache (Nervous system disorders) | 29 | 14
Neuropathy peripheral (Nervous system disorders) | 15 | 4
Insomnia (Psychiatric disorders) | 14 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 23

LIMITATIONS AND CAVEATS:
The study was terminated early due to business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the Sponsor for review. The Sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT05269355/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT05269355/SAP_001.pdf